CLINICAL TRIAL: NCT04437017
Title: Olanzapine or Dexamethasone, With 5-HT3 RA and NK-1 RA, to Prevent Nausea and Vomiting Induced by Cisplatin-Based Doublet Chemotherapy: A Non-inferiority, Prospective, Multi-Centered, Randomized, Controlled, Phase III Clinical Trial
Brief Title: Olanzapine or Dexamethasone, With 5-HT3 RA and NK-1 RA, to Prevent CINV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhigang Liu, Vice Director, Fifth Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No.ZDWY[2020]LunziNo.(K01-1)
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2021-05

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: nausea; vomiting; antiemesis
MeSH Terms: conditions — Vomiting; Nausea | interventions — Calcium Dobesilate; Fluprednisolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Olanzapine+NK-1 RA+5-HT3 RA (Experimental): Using one of the 5-HT3 receptor antagonists (a. Palonosetron: 0.25 mg d1 intravenous; b. Granisetron: 1 mg d1 intravenously, or 2 mg d1 orally; c. Ondansetron: 8-16 mg d1 intravenous or oral. the specific agent is chosen by the primary clinician, and is only delivered on the first day) within 30 minutes before cisplatin. Using one of the NK-1 receptor antagonists(a. Aprepitant: 125 mg orally, d1, 80 mg orally, d2-3; b. Fosaprepitant: 150 mg intravenously, d1) within 1 hour before cisplatin. On day 1-4, Olanzapine (5mg) is delivered orally after dinner.
  Interventions: Drug: Olanzapine+NK-1 RA+5-HT3 RA
- Dexamethasone+NK-1 RA+5-HT3 RA (Active Comparator): Using one of the 5-HT3 receptor antagonists (a. Palonosetron: 0.25 mg d1 intravenous; b. Granisetron: 1 mg d1 intravenously, or 2 mg d1 orally; c. Ondansetron: 8-16 mg d1 intravenous or oral. the specific agent is chosen by the primary clinician, and is only delivered on the first day) within 30 minutes before cisplatin. Using one of the NK-1 receptor antagonists (a. Aprepitant: 125 mg orally, d1, 80 mg orally, d2-3; b. Fosaprepitant: 150 mg intravenously, d1) within 1 hour before cisplatin. On first day, dexamethasone (12 mg) is given orally/intravenously within 30 minutes before cisplatin administered, and on day 2-4, the given dose of dexamethasone is 8 mg.
  Interventions: Drug: Dexamethasone+NK-1 RA+5-HT3 RA

INTERVENTIONS:
Drug: Olanzapine+NK-1 RA+5-HT3 RA — On day 1-4, Olanzapine (5mg) is delivered orally after dinner.
  Arms: Olanzapine+NK-1 RA+5-HT3 RA
Drug: Dexamethasone+NK-1 RA+5-HT3 RA — On first day, dexamethasone (12 mg) is given orally/intravenously within 30 minutes before cisplatin administrated, and on day 2-4, the given dose of dexamethasone is 8 mg.
  Other Names: Acidocont; Deronil; Dexacortal; Desameton; Fluprednisolone; (11β，16α）-9-Fluoro-11,17,21-trihydroxy-16-methylpregna-1,4-diene-3,20-dione
  Arms: Dexamethasone+NK-1 RA+5-HT3 RA

SUMMARY:
Chemotherapy-induced nausea and vomiting is a common side effect of cancer treatments, and dexamethasone offers a clear advantage over placebo for protection against chemotherapy-induced emesis in both acute and delayed phases. However, its side effects such as moderate to severe insomnia, hyperglycemia, dyspepsia, upper abdominal discomfort, irritability, increased appetite, weight gain and acne are gathering increasing concerns. Several clinical trials have shown that olanzapine plays an important role in treating delayed, refractory, breakthrough nausea and vomiting. Its side effects mainly include sedation and weight gaining. At present, the NCCN guidelines have recommended olanzapine-containing three-drug regimen for Highly Emetogenic Chemotherapy (HEC) and moderate emetic chemotherapy (MEC) to prevent vomiting, but its data in the Chinese population is limited. Hence, we initiated this prospective, multi-center, phase III study to validate the dexamethasone-free protocol: applying olanzapine to prevent CINV instead of dexamethasone.

ELIGIBILITY:
Inclusion Criteria (Patients are eligible to be included in the study only if they meet all of the following criteria):

1. Cancer patients, age ≥ 18 years and ≤75 years, ECOG score 0-2 points, receiving cisplatin-containing doublet chemotherapy such as cisplatin + gemcitabine / albumin paclitaxel / etoposide /fluorouracil / irinotecan / temozolomide as first line treatment;
2. Life expectancy ≥ 3 months;
3. Leucocytes≥3,000/uL;
4. AST≤2.5 × upper limit of normal;
5. Bilirubin ≤1.5 × upper limit of normal;
6. Serum creatinine ≤ 1.5 × upper limit of normal.

Exclusion Criteria (Patients will be excluded if any of the following criteria is met):

1. History of CNS disease, such as brain metastases or epilepsy;
2. Use of other antipsychotic drugs (such as risperidone, quetiapine, clozapine, phenothiazine, or butyrophenone, or such treatment is under scheduling during the study) within 30 days before enrollment; long-term use of phenothiazine as an antipsychotic agent;
3. Concurrent use of pharyngeal or abdominal radiotherapy;
4. Concurrent use of quinolone antibiotics;
5. Chronic alcoholism;
6. Known hypersensitivity to olanzapine;
7. Know arrhythmia, uncontrolled congestive heart failure or acute myocardial infarction within 6 months;
8. Known uncontrolled diabetes mellitus;
9. Vomiting or retching 24 hours before chemotherapy;
10. Use of anti-emesis drugs 48 hours before chemotherapy;
11. Concurrent use of amifostine;
12. Concurrent use of corticosteroids and the only anti-allergic choice is corticosteroids

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 557 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
0-120h Complete Remission Rate | 24 hours ,48 hours, 72 hours, 96 hours, 120 hours after chemotherapy
  The ratio of patients who have no vomiting and apply no anti-nausea drugs during the whole observation period.

SECONDARY OUTCOMES:
25-120 hours Complete Remission Rate | 24 hours , 48 hours, 72 hours, 96 hours, 120 hours after chemotherapy
  The ratio of patients who have no vomiting and apply no anti-nausea drugs during the 25-120 hours observation period.
0-120h No Nausea Rate | 24 hours, 48 hours, 72 hours, 96 hours, 120 hours after chemotherapy
  The ratio of patients who have no nausea during the whole observation period.

CONTACTS AND LOCATIONS:
Overall Officials: Zhigang Liu, M.D., Study Director — Fifth Affilliated Hospital of Sun Yat-sen University; Zhigang Liu, M.D., Principal Investigator — Fifth Affilliated Hospital of Sun Yat-sen University
Locations (1):
- Fifth Affilliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No